CLINICAL TRIAL: NCT06615856
Title: Understanding the Influence of Concomitant Irritable Bowel Syndrome (IBS) on Gastro-Oesophageal Reflux Disease (GORD), Including GORD-related Symptoms, GORD Severity, Oesophageal Motility, and Multi-Channel Intraluminal Impedance-pH Findings.
Brief Title: The Influence of Concomitant Irritable Bowel Syndrome on Gastro-Oesophageal Reflux Disease Symptoms and Severity.
Status: Not yet recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GA24/167199
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Irritable Bowel Syndrome; Gastro-oesophageal Reflux Disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastroesophageal Reflux | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients referred for high-resolution oesophageal manometry and multi-channel impedance pH testing: Patients that have been referred for high-resolution oesophageal manometry and multi-channel intraluminal impedance-pH monitoring at the Gastrointestinal Physiology department at Leeds Teaching Hospitals between September 2024 - January 2025 (subject to change based on recruitment time).
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Two questionnaires will be provided to participants to complete before their routine tests (which they would already be having regardless of the study and are not affected by their participation in the study).
  The questionnaires include: A Gastro-Oesophageal Reflux Symptom Questionnaire; and the ROME-IV Diagnostic IBS Module Questionnaire

SUMMARY:
This research aims to investigate whether there is a link between irritable bowel syndrome (IBS) and acid reflux, particularly whether there is a difference in acid reflux symptoms between people with and without IBS.

IBS is a functional gastrointestinal disorder, which has the same root cause as other functional gastrointestinal disorders that produce symptoms similar to acid reflux. Acid reflux symptoms may be typical (heartburn, regurgitation) or atypical (cough, sore throat, chest pain).

All participants are given two questionnaires: one to categorise them as either IBS or non-IBS, and one to understand their acid reflux symptoms. From this, the project will investigate whether there is a difference in the type (typical/atypical) and severity of acid reflux symptoms between people with and without IBS that attend for diagnostic acid reflux testing at Leeds Teaching Hospitals.

Two factors determine how much acid reflux someone has: the ability of the oesophagus (food- pipe) to move food from the throat to the stomach, and how well the muscle between the oesophagus and stomach works to keep acidic contents from moving back up.

All participants will have a test to see how well the muscles in their oesophagus are working. As there may be a link between IBS and oesophageal function, this project will investigate whether any patterns of abnormal oesophageal function can be identified in IBS patients that might explain their acid reflux symptoms.

Participants will then have a test that measures acid reflux over 24 hours, including the amount of acid and non-acid coming up, how high this reaches in the oesophagus, and whether symptoms are linked to these events.

Analysing these test results against questionnaire answers might help to understand the link between IBS and acid reflux to improve future diagnosis and treatment for the many people that have these conditions.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGIDs) are characterised by chronic gastrointestinal symptoms in the absence of demonstrable pathology, diagnosed using the Rome-IV criteria. IBS is the most prevalent FGID, affecting >12% UK population, accounting for 40-60% gastroenterology outpatient referrals. It is characterised by abdominal pain, bloating, and altered stool form or frequency, and is classified into four subtypes: IBS with predominant constipation; predominant diarrhoea; mixed bowel habits; or unsubtyped.

Whilst IBS pathogenesis is not wholly understood, it is considered attributable to visceral hypersensitivity (VH), disordered microbiota-brain-gut axis communication, gastrointestinal infection, and brain function changes. VH is an altered sensation response to physiological stimuli, which may occur from nervous system disturbances. Non-pathological visceral functions should not result in pain, yet the disordered response to physiological stimuli with VH causes an enhanced perception of mechanical triggers applied to the bowel, inducing perceived discomfort.

Oesophageal FGIDs with similar VH-mediated pathogenesis include functional heartburn (FH), reflux hypersensitivity (RH), functional chest pain, and globus. These can produce symptoms that are phenotypically indistinguishable from gastro-oesophageal reflux disease (GORD), yet exhibit no measurable cause.

GORD results from retrograde movement of acidic gastric contents into the oesophagus, characterised by excessive oesophageal acid exposure (OAE). Protective physiological mechanisms minimise gastro-oesophageal reflux, namely the anti-reflux barrier, comprising the lower oesophageal sphincter (LOS), crural diaphragm and supporting structures, along with peristaltic clearance of refluxate from the oesophagus. However, compromise of these mechanisms may cause gastro-oesophageal reflux to increase to pathological levels of OAE, resulting in oesophagitis and symptom generation.

Ambulatory pH-monitoring directly confirms or refutes GORD diagnoses by measuring OAE and reflux episode frequency over 24-hours. GORD can be classified as erosive reflux disease (ERD), diagnosed endoscopically by erosive oesophagitis or Barrett's oesophagus, or non-erosive reflux disease (NERD) which presents with no mucosal damage.

GORD can manifest diversely, with either typical or atypical symptoms. Typical symptoms include heartburn and acid regurgitation, whilst atypical manifestations include chest pain, chronic cough, belching, dyspepsia, globus, and more. Some studies have demonstrated that symptom presentation varies between ERD and NERD, with atypical symptoms presenting exceedingly in ERD, and typical manifestations more frequent with concurrent atypical symptoms.

NERD patients often report comparable symptom severity to ERD patients, despite typically conferring lower OAE, suggesting that clinically-relevant NERD may be concomitant with FGIDs or attributable to VH. Mechanoreceptor hypersensitivity may contribute to symptom perception, as one study found that those with NERD, FH and RH exhibited increased sensitivity to oesophageal balloon distension compared to controls and ERD patients. From this, it is hypothesised that predisposition to FGIDs may impact experienced GORD symptoms, regardless of OAE.

Previous studies have found significant overlap in the prevalence of GORD and IBS, suggesting shared underlying dysfunction. Furthermore, GORD concomitant with IBS has been found to present with exceedingly frequent atypical symptoms than GORD alone; however only a minority of symptoms were investigated, many of which may be specific to IBS. Additionally, males with IBS have been found to experience significantly greater reflux symptoms than controls, despite no GORD diagnoses, highlighting the potential influence of IBS on perceived symptoms. Moreover, IBS has been shown not to affect OAE, yet was associated with significantly higher GORD symptom scores, with influence comparable to OAE.

Whilst these studies demonstrate an association between IBS and GORD symptoms, the criteria that were used to diagnose IBS are outdated and oversimple, failing to distinguish between IBS subtypes. Furthermore, as the pH studies used measured only OAE to diagnose GORD, these are too simplistic to assess the potential influence of oesophageal FGIDs and non-acidic reflux on symptoms.

Improved understanding of the link between these conditions may enhance diagnosis and treatment for the abundance of people with both GORD and IBS. Therefore, this research primarily aims to investigate whether GORD concomitant with IBS manifests a particular presentation of symptoms, whether concomitance with IBS may influence GORD severity using multichannel intraluminal impedance-pH monitoring (MII-pH), and whether this differs between IBS subtypes.

MII-pH is the gold-standard for diagnosing GORD as it assesses weakly-acidic and non-acidic reflux, proximal extension, and baseline impedance, along with standard pH findings. It is essential for distinguishing NERD, RH and FH by classification of acid exposure time, non-acid reflux, and symptom association. Baseline impedance may also distinguish GORD and FH, as GORD has been shown to exhibit a lower baseline impedance due to reduced mucosal integrity. Furthermore, proximal reflux extension has been shown to correlate with atypical symptoms such as chronic cough, and is higher in those with NERD than RH, therefore is valuable for understanding symptom changes and distinguishing conditions. These previous findings necessitate the use of MII-pH in this project to wholly interpret any identifiable association between IBS and specific symptoms, by assessing the potential for a shared functional cause of IBS and oesophageal FGIDs. Therefore, this research further aims to investigate whether MII-pH parameters differ between IBS and non-IBS patients.

Additionally, a vague association has been identified between IBS and oesophageal motility, which may indicate that influence of IBS on GORD symptoms relates to smooth muscle dysfunction rather than functional causes. One study identified pathologically altered oesophageal motility patterns in IBS, while others found significantly lower LOS pressures, which may explain the overlap with upper gastrointestinal conditions. However, the significance of these findings in relation to the effect on GORD symptoms is unclear, particularly with the use of outdated conventional manometry to assess motility patterns and small sample sizes. Therefore, this project secondarily aims to investigate whether oesophageal motility patterns differ between IBS and non- IBS patients using high-resolution oesophageal manometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have been referred for high-resolution oesophageal manometry and ambulatory pH or multichannel intraluminal impedance-pH (MII-pH) studies at the Gastrointestinal Physiology department at Leeds Teaching Hospitals NHS Trust from September 2024 to January 2025 (dates subject to change depending on acquisition of approvals).
* All participants must be fully consenting with a good understanding of what the study involves.

Exclusion Criteria:

* Patients aged <18 years.
* Those that have not followed the pre-test preparation criteria, including: those that have not been sufficiently fasted prior to testing (6 hours for food, 3 hours for drinks); those that have not retained from taking proton pump inhibitor medication for 7 days prior to testing (lansoprazole, omeprazole, esomeprazole, rabeprazole, pantoprazole), histamine-2 receptor antagonist medication for 2 days prior to testing (famotidine, cimetidine, nizatidine), and other antacids on the day of testing (Gaviscon, Rennies, Peptac, etc).
* Patients that lack the capacity to understand, retain, and communicate information to accurately complete questionnaires relating to their experienced symptoms.
* Non-consenting patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential pool of participants includes those that have been routinely referred for high-resolution oesophageal manometry and ambulatory pH/multichannel intraluminal impedance-pH studies at the Gastrointestinal Physiology department at Leeds Teaching Hospitals NHS Trust from September 2024 to January 2025 (subject to change, depending on time of approval confirmation and recruitment time).
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2024-10-14 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
IBS Subtype | September 2024 - January 2025 (subject to change).
  Defined using the Rome-IV IBS module questionnaire, is necessary for grouping participants based on IBS symptoms and for building on previous research. The Rome-IV criteria is a well- established, verified tool for clinical diagnosis.
Gastro-oesophageal Reflux Symptoms | September 2024 - January 2025 (subject to change).
  The gastro-oesophageal reflux symptom questionnaire is suitable for assessing primary outcome measures of predominant symptom type, most bothersome symptom, and symptom severity. This is a valid for understanding participants' subjective perception of their symptoms and quantifies this with the use of closed questions.

SECONDARY OUTCOMES:
Gastro-Oesophageal Reflux Disease Severity | September 2024 - January 2025 (subject to change).
  Secondary outcome measures of acid exposure time and DeMeester score are well-established, objective measures of GORD severity.
Multi-Channel Intraluminal Impedance pH Findings | September 2024 - January 2025 (subject to change).
  Secondary outcome measures of baseline impedance, weakly acidic reflux, and proximal extent using multichannel intraluminal impedance-pH monitoring are valid and necessary for distinguishing gastro-oesophageal disorders.
High-Resolution Oesophageal Manometry Findings | September 2024 - January 2025 (subject to change).
  Secondary outcome measures of lower oesophageal sphincter resting pressure and % normal, weak, failed, spasmic, and hypertensive oesophageal contractions are valid for characterising oesophageal function, as per the standardised Chicago Classification protocol, obtained using gold-standard high-resolution oesophageal manometry.

IPD SHARING:
Plan to Share IPD: No
This research is for a Master's level project, with the purpose of assessing the students capability to conduct scientific research.